CLINICAL TRIAL: NCT02811783
Title: A Double Blind Randomized Vehicle Controlled Crossover Study to Evaluate the Safety and Efficacy of Topical Naloxone Hydrochloride Lotion 0.5% for the Relief of Pruritus in Patients With the MF or SS Forms of Cutaneous T-Cell Lymphoma
Brief Title: Naloxone Hydrochloride Study for Relief of Pruritus in Patients With MF or SS Forms of CTCL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Elorac, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EL-1007-01-01; 1R01FD005396-01A1 (FDA)
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Sézary Syndrome
Keywords: Pruritus; Mycosis Fungoides; CTCL; naloxone; opiate antagonist; Sézary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naloxone Hydrochloride Lotion, 0.5% (Active Comparator): Naloxone Hydrochloride Lotion 0.5%
  Interventions: Drug: Naloxone Hydrochloride Lotion, 0.5%
- Placebo Lotion (Placebo Comparator): Placebo Lotion
  Interventions: Drug: Placebo Lotion

INTERVENTIONS:
Drug: Naloxone Hydrochloride Lotion, 0.5% — Topical TID for 2 weeks
  Arms: Naloxone Hydrochloride Lotion, 0.5%
Drug: Placebo Lotion — Topical TID for 2 weeks
  Arms: Placebo Lotion

SUMMARY:
This multi-center, double-blind, vehicle-controlled, randomized crossover design study will evaluate the safety and efficacy of topically applied naloxone lotion, 0.5%, for the treatment of pruritus in patients with the mycosis fungoides (MF) or Sézary syndrome (SS) Forms of Cutaneous T-cell Lymphoma (CTCL). This study will also determine if there is systemic absorption of the drug in a subset of subjects and if so, describe the range and mean plasma levels reached after two weeks of three time daily (TID) dosing.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
There will be 160 subjects enrolled in the study. The study consists of a Screening Period of up to 7 days during which inclusion / exclusion criteria will be reviewed. Subjects meeting inclusion / exclusion criteria including the diagnostic criteria for MF or SS and a score of at least 5 on the 11-Point Numeric Rating Scale (NRS) for Pruritus will complete the one week Screening Period. Subjects will complete a daily diary for NRS for Pruritus scores and Sleep scores. At the end of the Screening Period, subjects who have a NRS for Pruritus score of at least 5 recorded in the diary on at least 4 of the 7 days preceding Day 0 will be eligible to continue. Baseline assessments will be recorded for vital signs, pruritic body surface area, skin integrity, PQOL, and laboratory results. The Baseline period will be followed by a 2 week Treatment Period 1 in which subjects will be randomized to Naloxone Lotion 0.5% or Placebo Lotion to be applied TID for 14 days. During the 2 week Treatment Period subjects will complete daily diaries of NRS for Pruritis scores and Sleep scores. On Day 14 subjects will return to the clinic to review diaries, adverse events (AEs), concomitant medications, and to record body surface area for pruritus, skin integrity, PQOL, and laboratory results. Subjects will then enter a Washout Period for up to 56 days until the subject again scores at least 5 on the NRS for Pruritus on 4 consecutive or 4 of the past 7 days or 56 days pass. Subjects will then enter a 2 week Treatment Period 2 during which the same procedures as Treatment Period 1 will be performed except subjects will receive the alternate treatment to that assigned in Treatment Period 1. Subjects will then have the option to enter a 26 Week Open Label Treatment Period 3 during which the same procedures as Treatment Period 1 and 2 will be performed except subjects will return only at Week 13 and Week 26 and all subjects will be treated with Naloxone Lotion 0.5%.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria for admission into the study:

1. Signed informed consent has been obtained.
2. Subject is at least 21 years of age.
3. Diagnosis of mycosis fungoides (MF) or Sézary syndrome (SS) will be based on a combination of histological, clinical, and immunophenotypical criteria. The histological criteria will be based on skin biopsy from the most representative skin area. The diagnostic criteria used for each subject will be specified in the case report forms and the specific classification of MF or SS will be identified. The TNMB system will be used to classify the stage of disease (See Section 8.4 for details).
4. Completion of the mSWAT assessment.
5. A history of pruritus that meets following criteria:

   At Screening Day -7:
   * present on a daily basis for greater than one month prior to Screening Day -7,
   * NRS for Pruritus score ≥5 as rated by the subject at the Day -7 Visit. Note: If the score is <5 and subject is taking or has taken a medication which may be affecting pruritus (e.g. systemic antihistamine or topical steroid), and if Investigator and subject agree, subject may washout or continue washout of medication and return for Day -7 Visit procedures after washout.

   At Baseline Period 1 Day 0:
   * NRS for Pruritus score of at least 5 recorded in the subject diary on at least 4 of the 7 days preceding Baseline Period 1 Day 0.
6. Pruritic treatment area of 5-95% of the subject's total treatable body surface area.
7. Subject can be expected to reliably follow treatment instructions and visit schedule.
8. Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, or intrauterine device) throughout the study or females of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year). A negative urine pregnancy test must be confirmed at Baseline screening for all female subjects who are not post-menopausal > 1 year or surgically sterile.
9. The subject agrees not to begin any new concomitant medications during their participation in the study, with the exception of medications necessary to treat infection, and to continue any concomitant medication throughout the study.
10. Subject has no visual or motor impairments that will make it difficult to complete the Daily Diary or apply the study medication.
11. Subject is able to speak, read, and write English and agrees to participate and comply with the study procedures.
12. Subject has a body mass index (BMI) between 18.5 and 30.5 kglm2 (see Appendix C, Body Mass Index Table) (subjects in PK subset only).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from study participation:

1. Pregnant or lactating female.
2. History of clinically significant heart failure.
3. Myocardial infarction within the past six months.
4. A history of ventricular arrhythmia requiring treatment.
5. Any medical condition which would, in the Investigator's opinion, preclude the subject from successfully participating in the study.
6. A known allergy to naloxone hydrochloride or any excipient in the formulation.
7. Previous naloxone use for pruritus.
8. Positive urine drug screen at Day 0 for opiates. Positive urine drug screen for anything other than opiates not explained, e.g., by concomitant medication, would also exclude the subject.
9. Treatment with any of the following during the restricted time period prior to Day -7, and at any time during the study, is not allowed:

Medication/Treatment Restriction:

Systemic narcotic analgesics (e.g. morphine, codeine) 7 days, Topical antihistamines to any skin surface [e.g. Zonalon® (doxepin)] 7 days, Other investigational drugs (excluding any therapies for the treatment of MF or SS) 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) for Pruritus | Baseline and 2 Weeks
  Change from Baseline to Day 14 in average NRS for Pruritus for each Treatment Period

SECONDARY OUTCOMES:
Responder Analysis - The difference in the proportion of subjects with a meaningful clinically significant improvement at the end of the two periods. | Baseline and 2 Weeks
  The difference in the proportion of subjects with a meaningful clinically significant improvement at the end of the two periods. A clinically significant improvement is defined as an improvement of at least one category on the 4-point (none, mild, moderate, severe) Likert Scale verbal rating scale (VRS) and at least two points on the 11-point NRS for Pruritus. The NRS for Pruritus scores will be converted to VRS scores as follows for the analysis: 0=none, 1-3=mild, 4-6=moderate, and 7-10=severe.
Numeric Rating Scale for Sleep | Baseline and 1 and 2 weeks
  The change from Baseline at each week of the NRS for Sleep average score for each Treatment Period.
Numeric Rating Scale for Pruritus | Baseline and 1 week
  The change from Baseline at Week 1 of the NRS for Pruritus average score for each Treatment Period.
Categorical Rating Scale (CRS) for Skin Integrity | Baseline and 2 weeks
  The change from Baseline at Week 2 of the CRS for Skin Integrity for each Treatment Period.
Pruritus Quality of Life Score (PQOL) | Baseline and Day 14 of each Treatment period
  The change from Baseline in the final categorization of the PQOL at Day 14 of each Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, MD, Study Director — Elorac, Inc.
Locations (16):
- United States (16):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Stanford University, Palo Alto, California
  - USSF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Cleveland Clinic Indian River Hospital, Vero Beach, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis University Dermatology, St Louis, Missouri
  - Washington University School of Medicine St. Louis, St Louis, Missouri
  - Stony Brook Dermatology, Stony Brook, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - University of Washington / Seattle Cancer Care Alliance (SCCA), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956